CLINICAL TRIAL: NCT01656122
Title: Pharmacokinetics of Abacavir Once Daily vs. Twice Daily and Lamivudine Once Daily vs. Twice Daily in HIV-infected Thai Children
Brief Title: Abacavir and Lamivudine PK in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Radboud University Medical Center (Other); amfAR, The Foundation for AIDS Research (Other); PHPT/AMS Laboratory, Faculty of Associated Medical Sciences, Chiang Mai University (Unknown); Chulalongkorn University (Other); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 167
Record Dates: First submitted 2012-07-17; First posted 2012-08-02 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: HIV
Keywords: pharmacokinetic paramters; abacavir; lamuvidine; HIV-infected children
MeSH Terms: interventions — abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PK (Experimental): PK of abacavir and lamivudine
  Interventions: Drug: abacavir; Drug: 3TC

INTERVENTIONS:
Drug: abacavir — Dosing of ABC will be according to the WHO guidelines by weight band for twice daily dosing. The once daily dosing will use the same mg/day as the twice daily dosing for that weight band
Drug: 3TC — Dosing of 3TC will be according to the WHO guidelines by weight band for twice daily dosing. The once-daily dosing will use the same mg/day as the twice-daily dosing for that weight band

SUMMARY:
The purpose of this study is to assess the pharmacokinetic parameters for ABC and 3TC in HIV-infected children younger than 18 years old with body weight ≥ 14 kgs.

DETAILED DESCRIPTION:
Abacavir (ABC) is a nucleoside reverse transcriptase inhibitor (NRTI) and continues to have good efficacy even in patients who have some resistant mutations to NRTIs. ABC is approved for use in children 3 months old and up. It is a preferred NRTI option for second line treatment in children in the World Health Organization guidelines (WHO). In the US and European guidelines, ABC is also recommended for first line treatment. Published studies support the efficacy and safety of twice and once daily ABC. In HIV-infected children < 12 years, ABC is licensed twice-daily only. However, ABC is licensed either twice-daily or once-daily for HIV-infected adults and children >12 years. In addition, ABC can be administered as the fixed dose combination once-daily with lamivudine (3TC), Kivexa, for HIV-infected adults and children >12 years.

Lamivudine (3TC) is a commonly used NRTI that is well tolerated and approved for young infants and children as a component in the first and second-line regimens in guidelines. Both once-daily and twice-daily 3TC are standard practice in many treatment guidelines although once-daily is US FDA-approved for age > 12 years only. The Thai Ministry of Health pediatric HIV treatment guideline recommend either once- or twice-daily as treatment options for children. The WHO currently recommends the twice-daily 3TC dosing only and encourages more pharmacokinetic studies of once-daily 3TC in children.

PK of ABC and 3TC in African and European children showed similar PK parameters for both twice daily and once daily dosing. There are no data on PK of ABC in Asian children and few studies on PK of 3TC in Thai children. Vanprapar et al. reported data in 42 Thai children weighing 6-30 kg participated in a cross-over PK study in which they received twice-daily dosing of generic fixed dose combination tablets of stavudine, 3TC, nevirapine or the liquid formulations of these drugs. The 3TC exposure was significantly higher with the tablet formulation but comparable to historical data in western adults and children taking branded tablets. Chokephaibulkit et al. reported higher 3TC exposure in 41 Thai HIV-infected children with 3TC tablets than 3TC solution.

There is strong evidence indicating that Asian patients, particularly Thais, have higher plasma concentrations for several ARVs compared to Westerners. Genetic differences between ethnicities may be the primary cause for altered drug metabolism, and as a result, different PK parameters. Higher drug concentrations in Thai adults have been shown for zidovudine, nevirapine, efavirenz, indinavir, lopinavir, atazanavir and saquinavir. Such high ARV concentrations were also shown in Thai children for nevirapine, indinavir, lopinavir and saquinavir. There are no data in Thai children for ABC. Only two studies evaluated 3TC concentration in Thai children using twice-daily dosing. It is conceivable that Thai children may have different PK profile of ABC and 3TC particularly once-daily dosing and than those reported in African and European children. In addition, using ABC and 3TC will provide an opportunity for Thai children to benefit from its once-daily dosing and good long-term safety particularly the favorable lipodystrophy and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of HIV infection using age-appropriate testing
2. Age < 18 years
3. Body weight ≥ 14 kgs
4. Currently treated with stable HAART within 30 days prior to enrollment
5. HIV RNA < 50 copies/ml
6. Have negative HLA B5701 or are currently on ABC-containing HAART and tolerating the regimen well
7. Caregivers give written informed consent and children aged 7 years and above who know their HIV status give assent

Exclusion Criteria:

1. Child/Caretaker refuse to participate in this study
2. Has vomiting or diarrhea > grade 3 (DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0 - December 2004, clarification dated August 2009) within 30 days prior to enrollment
3. Has the following laboratory toxicities > grade II according to the division of AIDS table for grading the severity of adult and pediatric adverse events within 30 days prior to enrollment:

   * SGPT
   * Hemoglobin
   * Creatinine
4. Has current active HIV-related infection
5. Has significant medical problem that would compromise the study results in the investigator's opinion
6. Pregnancy
7. Has history of poor adherence to ARV defined by less than 80% by pill count or by history within 30 days prior to enrollment
8. Concomitant treatment with drugs known to influence the PK of ABC (ribavirin, ethanol and methadone)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Ctrough and Area under the curve (AUC) of abacavir (ABC) and lamivudine (3TC) at week 2 and 4 | week 96
  assess the Ctrough and Area under the curve (AUC) of abacavir (ABC) and lamivudine (3TC) at week 2 twice daily dose and week 4 once daily dose

SECONDARY OUTCOMES:
CD4 | 96 weeks
  assess CD4 at weeks 48 and 96
viral load | 96 weeks
  assess viral load at weeks 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat Ananworanich, MD, PhD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok, Thailand

REFERENCES:
- [Result] Bunupuradah T, Punyahotra P, Cressey TR, Srimuan A, Thammajaruk N, Sophonphan J, Sriheara C, Burger DM, Puthanakit T, Ananworanich J. Plasma pharmacokinetics of once-daily abacavir- and lamivudine-containing regimens and week 96 efficacy in HIV-infected Thai children. J Virus Erad. 2015 Jul 1;1(3):185-91. doi: 10.1016/S2055-6640(20)30503-3. PMID 27482411
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org